CLINICAL TRIAL: NCT03941392
Title: Nutritional Study in Spanish Pediatric Population (EsNuPI)
Brief Title: Nutritional Study in Spanish Pediatric Population
Acronym: EsNuPI
Status: Completed | Type: Observational
Sponsor: Fundacion Iberoamericana de Nutricion (Other)
Collaborators: Universidad de Granada (Other); Fundación Española de la Nutrición (Other); CEU San Pablo University (Other); Lactalis (Industry)
Responsible Party: Sponsor
Other Study IDs: FF01/2019
Record Dates: First submitted 2019-04-22; First posted 2019-05-08 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Child, Only; Metabolic Diseases; Child Development; Diet Habit; Healthy Diet; Feeding Behavior; Health Behavior; Sedentary Lifestyle; Food Habits; Nutritional Status; Diet, Food and Nutrition
Keywords: Nutrition; Pediatric age; Physical activity; Dairy products; Dairy consumption; Sedentary habits; Diet quality; Children
MeSH Terms: conditions — Metabolic Diseases; Feeding Behavior; Health Behavior; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy children between 1 and 9 years old: A sample of 1500 apparently healthy children between 1 to 9 years old from urban areas from different regions of Spain.

SUMMARY:
This study investigates the aspects related to the intake of food and nutrients, physical activity and sedentary behavior of Spanish children from 1 to 9 years. Furthermore, the investigators will know if the consumption of dairy products is associated with a better dietary pattern.

Hypothesis: The habitual consumption of dairy products as part of a regular diet is associated with a better dietary pattern and a higher global diet quality.

DETAILED DESCRIPTION:
A prospective cross-sectional observational study in 1500 Spanish children (1 to 9 years) in urban areas >50,0000 inhabitants, distributed in eight regions (according to Nielsen Spanish areas) aiming to evaluate the food habits, dietary patterns, and nutrient intake, as well as physical activity behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between 1 and 9 years old without diseases carrying changes in the dietary patterns.
* Those following dietary advice such as for prevention of non-communicable chronic diseases

Exclusion Criteria:

* Children with any disease that cause changes in the dietary pattern and with any dietary restriction.
* Children suffering a metabolic disease such as hyperthyroidism or hypothyroidism.
* Children diagnosed with allergy and/or food intolerance like dairy allergy, milk allergy, lactose intolerance or cows milk protein allergy.
* Children with any chronic disease that causes changes in the dietary pattern
* Children who live in an institution (colleges, nursing homes, hospitals, host Institutions, etc )
* Children with a transitory pathology (flu, gastroenteritis, chicken pox, etc) at the time of the fieldwork.
* Children following a therapeutic diet due to recent surgery or any other medical prescription.
* Children related to Lactalis or Madison MK employees.
* Children whose parents or caregivers did not provide a signed consent form for their participation or not completed any study phase.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Apparently healthy children between 1 to 9 years who live in an urban area with more than 50 000 inhabitants in Spain and that answer all the study recalls
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Dietary habits | 10 months
  Dietary diversity and variety determinated by using a FFQ from last year of consumption, the FFQ consisted of 150 food items commonly used in the local Spanish cuisine. The FFQ asked about consumption of foods and beverages in portions per day, week or month
Food | 10 months
  Food groups will be obtained from the FFQ of last year's consumption, the FFQ consisted of 150 food items commonly used in the local Spanish cuisine. The FFQ asked about consumption of foods and beverages in portions per day, week or month. The food based dietary guidelines from Spain will be used to determine the number of portions consumed per food group.
Beverages | 10 months
  Beverage groups will be obtained from the FFQ of last year's consumption, the FFQ consisted of 150 food items commonly used in the local Spanish cuisine. The FFQ asked about consumption of foods and beverages in portions per day, week or month. The food based dietary guidelines from Spain will be used to determine the number of portions consumed per beverage group.
Energy, macro and micronutrient composition of the diet | 10 months
  Energy, macro and micronutrient composition of the diet determined by 2 24-h recalls
Active and sedentary habits | 10 months
  Active and sedentary habits were measured with the 1-week activity recall validated in children
Milk and dairy products consumption | 10 months
  Evaluate the different types of milk that children drink in 24 h, twice through 24 h dietary
Dietary quality index for children "KidMed" | 10 months
  Evaluate the quality of the diet through this quality index for the specific age group

SECONDARY OUTCOMES:
Growth and BMI | 1 year
  Determined by reported age, weight (kg), and height (cm)
Goldberg & Black cut-off for Energy Intake: Plausibility of the reported energy intake | 1 year
  Measured by the relation between the reported energy intake and the estimated energy expenditure. The cut-off points are determined by the information reported by the population itself.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Iberoamericana de Nutrición, Granada, Spain

IPD SHARING:
Plan to Share IPD: No